CLINICAL TRIAL: NCT04985487
Title: Regulatory Post-Marketing Surveillance (rPMS) Study for Brolucizumab(Beovu ® Injection, Beovu ®Prefilled Syringe)
Brief Title: Regulatory Post-Marketing Surveillance Study for Brolucizumab
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AKR01
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: nAMD; Neovascularized age related macular degeneration; Beovu; regulatory Post Marketing Study; Beovu Injection; Beovu Prefilled Syringe
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brolucizumab: Patients prescribed with brolucizumab in the approved indication
  Interventions: Other: brolucizumab

INTERVENTIONS:
Other: brolucizumab — Prospective observational study. There is no treatment allocation. Patients administered brolucizumab, that have started before inclusion of the patient into the study will be enrolled.
  Other Names: Beovu

SUMMARY:
This study is an open-label, multicenter, single-arm, observational post-marketing surveillance.

DETAILED DESCRIPTION:
The investigators will collect safety information and evaluate effectiveness in patients who are prescribed Beovu ® Injection, Beovu ®Prefilled Syringe (brolucizumab) in the approved indication after receiving informed consent over a period of 12 weeks. In addition, longer-term data (24 weeks, optionally 36 weeks) will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years with nAMD that are prescribed with Brolucizumab as per approved local product information
2. Patients who consent to participate in the study after the purpose and nature of the study have clearly explained to them (written informed consent)

Exclusion Criteria:

1. Contraindications as per local prescribing information 1) Hypersensitivity to the active substance or to any of the excipients. 2) Active or suspected ocular or periocular infection. 3) Active intraocular inflammation.
2. Patients participating in other investigational drug trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years who present to the participating study sites, where the decision to newly prescribe Beovu ® Injection, Beovu ®Prefilled Syringe (brolucizumab) were made prior to evaluating eligibility for this study.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events at 12 weeks | 12 weeks
  Incidence of adverse events and serious adverse events

SECONDARY OUTCOMES:
Incidence of adverse events at 24 weeks and optionally at 36 weeks | Up to 36 weeks
  Incidence of adverse events and serious adverse events
Proportion of patients gaining or losing more than 15 letters on the ETDRS chart | Week 12, week 24, optionally week 36
  The ETDRS chart has been introduced as a standardized visual acuity (VA) testing chart. It uses 14 lines of 5 Sloan letter optotypes in each line in logarithmic progression. The space between lines and letters is proportionally equal keeping the effect of contour interaction constant. The threshold VA corresponds to the line in which 3 out of 5 optotypes were correctly identified. Alternatively, a by-letter scoring system (-0.02 logMAR credited for each letter correctly read) can be used. The testing distance can be varied; the corresponding visual acuity can be read easily from the chart. The chart is mounted on a box that is backlit by fluorescent tubes. For repeated measurements, the chart itself can be exchanged, providing different letters for different eyes.
Mean change of Central Subfield Thickness (CST) from baseline | Baseline, week 12, week 24, optionally week 36
  CST is measured as one parameter by Optical coherence tomography.
Mean change of Best Corrected Visual Acuity (BCVA) from baseline | Baseline, week 12, week 24, optionally week 36
  BCVA is the best possible vision that an eye can achieve with the use of glasses or contact lenses. It is measured by ETDRS chart or equivalent with the use of glasses or contact lenses
Mean Best Corrected Visual Acuity (BCVA) | Baseline, week 12, week 24, optionally week 36
  BCVA is the best possible vision that an eye can achieve with the use of glasses or contact lenses. It is measured by ETDRS chart or equivalent with the use of glasses or contact lenses
Mean Central Subfield Thickness (CST) | Baseline, Week 12, week 24, optionally week 36
  CST is measured as one parameter by Optical coherence tomography.
Number of injections | Up to 36 weeks
  Number of Brolucizumab injections to be collected
Percentage of patients completing the loading phase | 4 months
  Loading phase: ≥ 3 injection during first 4 months
Percentage of patients who maintained with 12 weeks interval | Up to 36 weeks
  Percentage(%) of patients who maintained with 12 weeks interval
Proportion of patients with retinal fluid | Week 12, week 24, optionally week 36
  Proportion of patients with Intraretinal fluid (IRF), subretinal fluid (SRF) or sub-retinal pigment epithelium (sub-RPE) fluid defined as presence/absence
Prior anti-VEGF treatment history - number of prior injections | Baseline
  Number of injections of prior anti- vascular endothelial growth factor (VEGF) treatment
Prior anti-VEGF treatment history - agent of prior injections | Baseline
  Agent of prior anti - vascular endothelial growth factor (VEGF) injections
Predictive factors of treatment outcomes (persistent disease activity) | Week 24
  Predictive factors of patients identified with persistent disease activity. Persistent disease activity is defined as presence of fluid and CST of at least 200µm
Treatment naïve/non-naïve | Baseline
  Number of participants that are treatment naïve / non-naïve to be collected
Treatment interval | Up to week 36
  Number of participants by treatment interval to be collected
Concomitant treatments | Baseline
  Number of participants with concomitant treatments to be collected
Number of participants with post injection empirical treatment | Week 12, week 24, optionally week 36
  Post injection emperical treatment means any medication or therapy (usually topical medication such as topical antibiotics, topical steroid..etc.) routinely prescribed on the same day of injection in order to prevent post injection complications. It is differentiated from concomitant medication.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- South Korea (14):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Goyang-si, Gyeonggi-do
  - Novartis Investigative Site, Guri-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Iksan Si, Jeonlabuk Do
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Jeju City
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu

IPD SHARING:
Plan to Share IPD: No